CLINICAL TRIAL: NCT00178230
Title: Circulating Cytokines as Predictors of Radiation Induced Pulmonary Toxicity in Thoracic Malignancies
Brief Title: Circulating Cytokines as Predictors of Radiation Induced Pulmonary Toxicity
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Yuhchyau Chen, Proffessor, University of Rochester
Other Study IDs: URCC 4595
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is being conducted by the University of Rochester Cancer Center to determine the levels of cytokines in the blood, and to determine if blood levels of these cytokines are related to the side effects of radiation therapy combined with other treatments.

ELIGIBILITY:
Inclusion Criteria:

Patients receiving radiation therapy for lung cancer combined with surgery either pre or post RT to the chest for lung cancer not associated with atelectasis, pleural effusion.

Patients receiving HDR Brachytherapy for lung cancer.

Patients receiving concomitant radiation and interferon therapy for lung cancer.

Patients receiving concomitant chemotherapy and radiation for lung cancer. Prior drug therapy does not make patients ineligible.

Karnofsky ≥ 70 %.

There are no age restrictions.

Acceptable bone marrow function - WBC 2 3000/mm3, platelet count > 100,000, hematocrit ≥ 33%, hemoglobin ≥ 11 gms/dl.

Life expectancy > 6 months.

Patients must sign informed consent meeting all federal and institutional guidelines.

Exclusion Criteria:

Patients not meeting eligibility criteria stated above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving radiation therapy for lung cancer combined with surgery either pre or post RT to the chest for lung cancer not associated with atelectasis, pleural effusion.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 1996-03-15 (Actual); Primary Completion 2013-11-25 (Actual); Study Completion 2013-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuhchyau Chen, MD, Ph.D, Principal Investigator — Universtiy of Rochester, Dept of Radiation Oncology
Locations (1):
- University of Rochester, Dept. Radiation Oncology, Rochester, New York, United States